CLINICAL TRIAL: NCT05894707
Title: A Randomized, Double-blinded, Dose-escalation Phase Ia Study to Evaluate the Safety and Tolerability of SCT650C in Healthy Volunteers
Brief Title: Evaluate the Safety and Tolerability of SCT650C in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SCT650C-612-1-01
Record Dates: First submitted 2023-05-29; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Autoimmune Disease
Keywords: IL-17A monoclonal antibody
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 80 mg SCT650C or normal saline (Experimental): Eight qualified participants will be randomized at a ratio of 6:2 to receive 80 mg SCT650C or normal saline on Day 1
  Interventions: Drug: SCT650C
- 160 mg SCT650C or normal saline (Experimental): Eight qualified participants will be randomized at a ratio of 6:2 to receive 160 mg SCT650C or normal saline on Day 1
  Interventions: Drug: SCT650C
- 40 mg SCT650C or normal saline (Experimental): Eight qualified participants will be randomized at a ratio of 6:2 to receive 40 mg SCT650C or normal saline on Day 1
  Interventions: Drug: SCT650C
- 20 mg SCT650C or normal saline (Experimental): Eight qualified participants will be randomized at a ratio of 6:2 to receive 20mg SCT650C or normal saline on Day 1
  Interventions: Drug: SCT650C

INTERVENTIONS:
Drug: SCT650C — Recombinant anti-IL-17A antibody
  Other Names: Recombinant anti-IL-17A antibody

SUMMARY:
The goal of clinical trial is to evaluate the safety and tolerability of SCT650C in healthy participants.

DETAILED DESCRIPTION:
Interleukin-17A (IL-17A) is a new potential therapeutic target which plays important role in pathogenesis of several autoimmune disorders including psoriasis, rheumatoid arthritis, possibly - systemic lupus erythematosus (SLE) and multiple sclerosis (MS). SCT650C is a novel humanized monoclonal antibody against human IL-17A developed by Sinocelltech which is now on the first step of clinical evaluation. SCT650C-612-1-01 study is the first-in-human clinical trial which is intended to evaluate tolerability, safety, pharmacokinetics and immunogenicity of SCT650C in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 18 to 65 years, inclusive, at the time of screening; 1a) Women of childbearing potential (WOCBP) must have a negative serum pregnancy test at screening and a negative urine pregnancy test at Day -1 and must not be breastfeeding, lactating or planning pregnancy during the study period. WOCBP must maintain an acceptable form of contraception (see Appendix 2) from Screening until 180 days from study drug dosing;

   • WOCBP are defined as any female who has experienced menarche, who has not undergone surgical sterilization (hysterectomy, bilateral oophorectomy, bilateral salpingectomy or tubal ligation) and is not postmenopausal;
   * Menopause is defined as 12 months of amenorrhea in the absence of other biological causes. This will be confirmed by documented serum follicle stimulating hormone (FSH) levels > 40 milli-International unit/mL to confirm menopause;
   * Contraception requirements do not apply to WOCBP in same-sex relationships. 1b) A male subject with a female partner of childbearing potential is eligible to participate if he agrees to use acceptable contraception (see Appendix 2) during the treatment period and for at least 180 days post dose.
   * Contraception requirements do not apply to:

     - male participants in same-sex relationships, or

     - male participant whose female partners are not of childbearing potential, whether surgically sterile or postmenopausal (FSH level required).
   * Male participants should avoid donating sperm for at least 180 days post-dose.
2. Healthy male and female participants, with no significant medical history, and in good health as determined by detailed medical history, full physical examination, vital signs, 12-lead electrocardiogram (ECG), and laboratory tests;
3. Body mass index (BMI) 18-32 kg/m2 and male weight ≥50 kg, and female weight ≥45 kg during the screening;
4. Participants who signed the informed consent, and are considered reliable and capable of adhering to the protocol (e.g., able to understand), visit schedule, and medication intake according to the judgment of the investigator.

Exclusion Criteria:

* 1) Recent use of any biological agents within 3 months before screening. Biological agents encompass a range of medicines derived from biological sources, including but not limited to some vaccines, growth factors, immune modulators, monoclonal antibodies, and products derived from human blood and plasma.

  2) Recent use of prescription medicines, over-the-counter medicines, vitamins or supplements within 7 days, or 5 half-lives (whichever is longer) prior to dosing at the investigators' discretion.

  3) Vaccination with live vaccine within 4 weeks prior to study drug administration, vaccination with an inactivated vaccination within 2 weeks prior to study drug administration, or intention to receive a live vaccine during the study period.

  4) Participants who have received an investigational drug in the previous 90 days or 5 half-lives, whichever is longer, prior to Day 1 dosing.

  5) Participants have a known allergy or hypersensitivity to any biologic therapy that would pose an unacceptable risk to the participant if participating in this study.

  6) Acute infection within 30 days prior to study drug administration. 7) Participants with active tuberculosis or latent tuberculosis, or those with history of previous tuberculosis infection.

  8) Histories of lymphoproliferative disease within 5 years; current history of malignancy or a history of malignancy within 5 years (except for squamous cell carcinoma of the skin, basal cell carcinoma, and cervical cancer in situ after thorough treatment without any signs of recurrence).

  9) Participants with a personal history of, or symptoms consistent with, inflammatory bowel disease (IBD).

  10) Associated with an active infection, or with an infection history: a. Systemic anti-infective treatment 4 weeks before administration of study drug; b. Serious infection with hospitalization or intravenous anti-infective treatment within 8 weeks before administration of study drug; c. Recurrent, chronic or other active infections, which are assessed by the investigator to increase the risk of the participant.

  11) Positive results of any of the following: Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (HBcAb), Hepatitis B virus (HBV) deoxyribonucleic acid (DNA), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody, interferon-gamma release assay (IGRA) or treponema pallidum particle agglutination (TPPA).

  12) Female participants who are breastfeeding, pregnant, or male participants who plan to father children during the study.

  13) Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels >1.5 times the upper limit of normal (ULN) at screening or Day -1; White cell count < 3.0; Neutrophil count < 2.0; Platelet count < 150. These tests can be repeated once at the investigator's discretion 14) Presence of any medical condition, mental health condition or suicidal ideation/behavior, which would make the participant unsuitable for inclusion in the study.

  15) Participants who underwent major surgery within 8 weeks prior to baseline, or are planning to undergo major surgery during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Baseline (Day 1, IP administration) up to 24 weeks
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

SECONDARY OUTCOMES:
Percentage of participants with at least one treatment-emergent serious adverse event (SAE) | Baseline (Day 1, IP administration) up to 24 weeks
  An SAE is any AE that fulfills one or more of the following:
  * Results in death;
  * Is life-threatening;
  * Requires hospitalization or prolongation of existing hospitalization;
  * Results in persistent or significant disability or incapacity;
  * Results in a congenital abnormality or birth defect;
  * Important medical event
Peak Plasma Concentration (Cmax) of SCT650C | Baseline (Day -1 predose) up to 24 weeks
  Pharmacokinetics: Cmax is the maximum observed concentration of SCT650C into serum.
Area under the plasma concentration versus time curve (AUC) of SCT650C | Baseline (Day -1 predose) up to 24 weeks
  Pharmacokinetics: Area Under the Concentration Versus Time Curve (AUC) from time zero to infinity was reported.
The level of anti-drug antibodies (ADA) to SCT650C | Baseline (Day -1 predose) up to 24 weeks
  Immunogenicity as measured by anti-drug antibodies (ADA) to SCT650C over time

CONTACTS AND LOCATIONS:
Overall Officials: Sam Salman, Principal Investigator — Linear Clinical Research
Locations (3):
- Australia (3):
  - Linear Clinical Research - Joonadalup, Joondalup, Western Australia
  - Linear Clinical Research - B Block, Nedlands, Western Australia
  - Linear Clinical Research - Harry Perkins, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No